CLINICAL TRIAL: NCT04130204
Title: Randomized, Double-blinded, Placebo-controlled Study of the Efficacy and Safety of DYV700 for Reducing Pain Associated With an Acute Gout Flare
Brief Title: Topical Application to Relieve Gout: Efficacy Trial & Safety (TARGETS)
Acronym: TARGETS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dyve Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DYV-702
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Topical lotion is provided in de-identified sachets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): DYV700, 10mL 3 times per day for 7 days Colchicine 1.2mg plus 0.6 mg 1 hour later at onset of flare (SOC)
  Interventions: Drug: DYV700; Drug: Colchicine 0.6 mg
- Placebo (Placebo Comparator): Placebo, 10mL 3 times per day for 7 days Colchicine 1.2mg plus 0.6 mg 1 hour later at onset of flare (SOC)
  Interventions: Drug: Placebo; Drug: Colchicine 0.6 mg

INTERVENTIONS:
Drug: DYV700 — Proprietary transdermal delivery platform
  Arms: Active
Drug: Placebo — Vehicle transdermal delivery platform
  Arms: Placebo
Drug: Colchicine 0.6 mg — Standard of care, 2 tablets (1.2 mg) loading dose followed by 1 tablet (0.6 mg) 1 hour later at onset of gout flare.

SUMMARY:
This overall goal of this trial will be to demonstrate that DYV700 is safe and effective as a treatment for acute gout flares.

DETAILED DESCRIPTION:
Gout presents as intermittent acute painful and debilitating gout flares. High serum uric acid levels lead to the deposition of urate crystals in and around the joints, most commonly the big toe (also called podagra) and other peripheral joints. An acute gout flare causes extreme pain and inflammation of the afflicted joints. It initially presents as a monoarticular condition but can affect several joints as the disease progresses. Gout flares typically take 7-10 days to resolve.

Currently, the inflammation and pain associated with acute gout flares are treated anti-inflammatories, including non steroidal anti-inflammatory drugs (NSAIDs), colchicine, corticosteroids, and adrenocorticotropic hormone. However these drugs are limited in efficacy, contraindicated for some patients and may take more than 24 hours to relieve gout symptoms (e.g. colchicine).

DYV700 will be developed to reduce the pain associated with acute gout flares. DYV700 is applied topically and utilizes a proprietary drug delivery system to deliver it's active ingredients.

ELIGIBILITY:
Key Inclusion Criteria:

1. Females and males, age 18 to 75 years of age.
2. Diagnosis of gout using ACR/EULAR criteria (must have a score of equal to or greater than 8)
3. Subjects must have experienced ≥2 gout flares in the 12 months prior to screening;
4. Subjects that have not changed their urate lowering therapy (ULT) in the 2 weeks prior to the start of the gout flare and who will remain on the same dose throughout the follow-up period of the trial.
5. If taking NSAID, oral steroids, opioids, or other pain medications at standard doses (as stated on drug label) for pain unrelated to their gout flare, must be taking the same drug for at least 7 days prior to the gout flare and throughout the length of the trial.
6. Women of childbearing potential are excluded. Women not considered of childbearing potential must have one of the following documented in their study medical history:

   1. Postmenopausal for at least 12 months prior to study;
   2. Without a uterus and/or both ovaries; or
   3. Bilateral tubal ligation at least six months prior to study enrollment.

Key Exclusion Criteria:

1. BMI of >40kg/m2 at the time of screening
2. Subjects that have not changed their urate lowering therapy (ULT) in the 2 weeks prior to the start of the gout flare and who will remain on the same dose throughout the follow-up period of the trial.
3. Subjects who are contraindicated for the use of colchicine or whom are unable to take the SOC dose of 1.2mg followed by 0.6mg an hour later.
4. Subjects with rheumatoid arthritis, psoriatic arthritis, evidence/suspicion of infectious/septic arthritis, acute polyarticular gout (4 or more joints), with arthritis due to any cause other than gout that may confound any study assessments per Investigator discretion.
5. Subjects who have experienced >2 gout flares per month, or >12 attacks overall in the months prior to randomization.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Pain Intensity in the Target Joint | Baseline-7 days
  Sum of pain intensity differences (SPID) from baseline to Day 7 in the target joint, using a 11-point (0-10) numeric rating scale (NRS) pain scale with 0-No Pain and 10-The Most Intense Pain Imaginable

SECONDARY OUTCOMES:
Time to Resolution | Baseline-7 days
  Time to resolution (with resolution defined as a ≥ 50% reduction in target joint pain score from baseline)
Rescue Medication Usage | Baseline-7 days
  Usage of rescue medications for pain throughout treatment period
Swelling | 24 hours and 7 days
  Swelling of the target joint as rated by a clinician using a Likert Scale 0- No swelling
  1- mild swelling, 2- moderate swelling, 3- severe swelling (or bulging beyond joint margins)
Tenderness | 24 hours and 7 days
  Tenderness of the target joint as rated by a clinician using a Likert Scale 0= Patient States "no pain", 1= Patient states "there is pain and winces", 2= Patient states "there is pain, winces and withdraws"
PROMIS PF 20 | Baseline (prior to product application and colchicine use), day 2 and day 7
  Physical Function Questionnaire
Level of Improvement | 24 hours, day 2 and day 7
  Subject Reported Assessment of Improvement Likert Scale 0= excellent, 1= very good, 2= good, 3= fair, 4= poor response to treatment

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline-7 days
  Adverse event and serious adverse event incidence during trial period

CONTACTS AND LOCATIONS:
Locations (1):
- Smitha Reddy, Poway, California, United States

IPD SHARING:
Plan to Share IPD: No